CLINICAL TRIAL: NCT06801652
Title: The Influence of Sperm Morphology and Functional Indices on Blastocyst Development in Assisted Reproduction
Status: Completed | Type: Observational
Sponsor: Calla IVF Center (Other)
Responsible Party: Sponsor
Other Study IDs: CALLA TERATOZOOSPERMIA
Record Dates: First submitted 2025-01-25; First posted 2025-01-30 (Actual); Last update posted 2025-01-30 (Actual); Status verified 2025-01

CONDITIONS: Spermatozoa, Abnormal; in Vitro Fertilization; Blastocyst; Aneuploidy
MeSH Terms: conditions — Teratozoospermia; Aneuploidy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Positive HCG pregnancy test after embryotransfer: Patients with sperm morphology indexes analyzed and had at least one good quality blastocyst that had a Positive HCG pregnancy test after embryo-transfer.
  Interventions: Other: Sperm morphology indexes
- Negative HCG pregnancy test after embryotransfer: Patients with sperm morphology indexes analyzed and had at least one good quality blastocyst that had a Negative HCG pregnancy test after embryo-transfer.
  Interventions: Other: Sperm morphology indexes
- No embryo obtained after IVF: Patients with sperm morphology indexes analyzed and had no blastocyst in day 5 or 6 after ICSI-IVF.
  Interventions: Other: Sperm morphology indexes
- All embryos obtained are aneuploid: Patients with sperm morphology indexes analyzed and had all blastocyst of day 5/6 tested and aneuployd after ICSI-IVF.
  Interventions: Other: Sperm morphology indexes

INTERVENTIONS:
Other: Sperm morphology indexes — We analyzed all sperm morphology indexes in all groups.

SUMMARY:
Samples from male partners of 120 infertile couples undergoing IVF were analyzed. Sperm morphology was assessed using the SpermBlue staining method, while TZI, MAI, and SDI were calculated. Embryo development was monitored until day 5 or 6. Statistical analyses included regression models and correlation coefficients to evaluate the predictive value of sperm indices on blastocyst development.

DETAILED DESCRIPTION:
For spermatozoa selection we used ZyMot multi in all patients undergoing IVF. After intracytoplasmatic injection of spermatozoa we asses the blastocyst grading in day 5. NEQSI score meaning numerical embryonic quality score index was used for statistical purpose. The spermatozoa morphology indexes were: TZI (teratozoospermia index), MAI (multiple anomalies index), SDI (sperm deformity index) and analyzed with CASA analyzer. All these indexes were assessed in patients and correlated in all groups: patients that had a positive pregnancy test, patients that had a negative pregnancy rate, patients that had no blastocyst in day 5 and patients that had all aneuploid embyos.

ELIGIBILITY:
Inclusion Criteria:

* couples with an infertility diagnosis that underwent an IVF procedure and had obtained at least one blastocyst

Exclusion Criteria:

* donors
* uterine abnormalities

Ages: 21 Years to 40 Years | Sex: All
Age Groups: Adult
Study Population: This prospective observational study analyzed sperm and embryonic parameters from 120 IVF cycles over 18 months. Functional sperm indices and embryo outcomes were evaluated to determine their relationship.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2023-10-21 (Actual); Primary Completion 2024-10-23 (Actual); Study Completion 2024-11-10 (Actual)

PRIMARY OUTCOMES:
Evaluation of sperm morphology indices on fertilization and blastulation rate | 18 months
  Functional sperm indices and embryo outcomes were evaluated to determine their relationship.

SECONDARY OUTCOMES:
Evaluation of sperm morphology indices on IVF outcomes | 16 months
  The study's findings are limited to IVF populations and may not generalize to natural conception.

CONTACTS AND LOCATIONS:
Locations (1):
- Calla Ivf Center, Oradea, Bihor County, Romania